CLINICAL TRIAL: NCT05097547
Title: Contingency Management for Stimulant Use Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Nassima Ait-Daoud Tiouririne, Principal Investigator, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSR210335; 17803 (Other: HSR Submission Number)
Record Dates: First submitted 2021-10-01; First posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Stimulant Use; Contingency Management

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Contingency management (Experimental): This arm will include data from participants who received CM
  Interventions: Behavioral: Contingency Management

INTERVENTIONS:
Behavioral: Contingency Management — Contingency management involves receiving monetary prizes in exchange for negative urine drug screens.

SUMMARY:
The invetigators' objective is to implement Medication Assisted Treatment (MAT) and contingency management in patients affected by co-occurring opioid use disorder and stimulant use disorder. Participants will continue to receive standard of care for their opioid use disorder via MAT at our Outpatient Based Opioid Treatment (OBOT) Clinic. Participants' stimulant use disorder will be targeted through contingency management, with twice weekly urine drug screens and monetary prizes in exchange for negative urine drug screens. Through regular clinic visits and the use of incentives, the investigators hope to increase treatment adherence and increase the number of negative urine drug screens in subjects struggling with co-morbid opioid use disorder and stimulant use disorder. The investigators will determine whether or not this treatment is effective in this population, versus conventional treatment (baseline therapy patients were getting through OBOT). The investigators' primary outcome measure will be stimulant abstinence duration during the twelve week study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Patients treated for opioid use disorder in the Outpatient Based Opioid Treatment (OBOT) Clinic and who also struggle with stimulant use disorder but failed conventional treatment (positive urine drug screen for substances other than THC and buprenorphine)
* Ideal candidates will test positive for 3 out of 4 weeks or more prior to starting contingency management

Exclusion Criteria:

* Persons under the age of 18
* Persons not able to attend follow-up clinic visits
* Persons not able to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
stimulant abstinence | 12 weeks
  Duration of stimulant abstinence based on urine drug screens

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ginley MK, Pfund RA, Rash CJ, Zajac K. Long-term efficacy of contingency management treatment based on objective indicators of abstinence from illicit substance use up to 1 year following treatment: A meta-analysis. J Consult Clin Psychol. 2021 Jan;89(1):58-71. doi: 10.1037/ccp0000552. PMID 33507776
- [Result] McPherson SM, Burduli E, Smith CL, Herron J, Oluwoye O, Hirchak K, Orr MF, McDonell MG, Roll JM. A review of contingency management for the treatment of substance-use disorders: adaptation for underserved populations, use of experimental technologies, and personalized optimization strategies. Subst Abuse Rehabil. 2018 Aug 13;9:43-57. doi: 10.2147/SAR.S138439. eCollection 2018. PMID 30147392
- [Result] Miguel AQ, Madruga CS, Cogo-Moreira H, Yamauchi R, Simoes V, da Silva CJ, McPherson S, Roll JM, Laranjeira RR. Contingency management is effective in promoting abstinence and retention in treatment among crack cocaine users in Brazil: A randomized controlled trial. Psychol Addict Behav. 2016 Aug;30(5):536-543. doi: 10.1037/adb0000192. Epub 2016 Jul 21. PMID 27442691